CLINICAL TRIAL: NCT05504018
Title: Clinical and Radiological Evaluation of Anterior Cruciate Ligament Reconstruction Surgery With Follow-up at Least 1 Year
Brief Title: Clinical and Radiological Evaluation of ACL Reconstruction Results
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsun University (Other)
Responsible Party: Principal Investigator, Ahmet Emin Okutan, Specialist in Orthopaedics, Samsun University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: AEOACL
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Anterior Cruciate Ligament Injuries
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: ACL reconstruction — Anterior cruciate ligament reconstruction surgery

SUMMARY:
The study is intended to include all patients who will undergo surgical reconstruction of the anterior cruciate ligament (ACL). The patients will be monitored and evaluated preoperatively and also at 6 months and 1 years after the intervention through a clinical visit. Such assessments will include the patient reported outcomes, the objective examination of the knee during a medical examination to quantify its stability and the radiological examination.

DETAILED DESCRIPTION:
The literature presents a number of studies on the reconstruction of the anterior cruciate ligament, as well as numerous registers, but the identification of factors and parameters determining the outcomes remains largely debated. The study aims to analyze the potentially individual and operative parameters and identify the factors responsible for the clinical and radiological outcomes. In addition to collecting patient data in terms of features and clinical-radiological status, objective data will be documented and correlated.

The study is intended to include all patients who will undergo surgical reconstruction of the anterior cruciate ligament (ACL). These patients will be followed and evaluated preoperatively, at 6 months and at 1 years after surgery during a clinical visit. Such assessments will include the patient reported outcomes, the objective examination of the knee during a medical examination to quantify its stability and the radiological examination.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have provided informed written written consent;
* Patients aged between 18 and 45;;
* Patients undergoing reconstructive surgical treatment of the anterior cruciate ligament (ACL)

Exclusion Criteria:

* Patients who have not signed informed consent;
* Patients undergoing any additional concomitant ligament repair or reconstruction at the same surgery
* Revision procedures
* Patients unable to lay still in an MRI or CT scanner
* Patients with a torn ACL or previous ACL reconstruction in the contralateral knee.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-02 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Magnetic Resonance Imaging (MRI) of Graft | 1 year
  Graft maturation on MRI using T2 Turbo Spin Echo (TSE) sequence without fat saturation

SECONDARY OUTCOMES:
Difference in Computed Tomography (CT) imaging of Tunnels | 1 day, 6 months, 1 year
  Femoral and Tibial Tunnel Morphological Changes
International Knee Documentation Committee (IKDC) | 1 year
  Patient reported outcome measures of symptoms, sports activity & knee function. 0-100 points with 0 (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms)
Marx Activity Rating Score | 1 year
  Clinical Outcomes
Isokinetic Dynamometer | 1 year
  Measurement of knee extension and flexion torque using the isokinetic dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Emin Okutan, MD, Principal Investigator — Samsun University
Locations (1):
- Ahmet E. Okutan, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Putnis SE, Klasan A, Oshima T, Grasso S, Neri T, Coolican MRJ, Fritsch BA, Parker DA. Magnetic Resonance Imaging Assessment of Hamstring Graft Healing and Integration 1 and Minimum 2 Years after ACL Reconstruction. Am J Sports Med. 2022 Jul;50(8):2102-2110. doi: 10.1177/03635465221096672. Epub 2022 May 25. PMID 35612835